CLINICAL TRIAL: NCT07168655
Title: Real-World Patients With Obstructive Hypertrophic Cardiomyopathy Treated With Mavacamten - a Single-Center Descriptive Study
Brief Title: Mavacamten in Obstructive Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1039
Record Dates: First submitted 2025-07-23; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy (oHCM)
Keywords: Obstructive Hypertrophic cardiomyopathy (oHCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants prescribed mavacamten treatment
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — According to the product label

SUMMARY:
The purpose of this study is to evaluate the real-world outcomes of individuals diagnosed with obstructive hypertrophic cardiomyopathy (oHCM) treated with mavacamten at the Hospital of The University of Pennsylvania in the US

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at index date
* Prescription of mavacamten for the treatment of Obstructive Hypertrophic Cardiomyopathy (oHCM)
* ≥ 4 weeks of follow-up after prescription of mavacamten

Exclusion Criteria:

* Data collection as part of a clinical trial during the study period
* Current participation in a myosin inhibitor clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of adult individuals diagnosed with Obstructive Hypertrophic cardiomyopathy (oHCM) that have been prescribed mavacamten at The Hospital of the University of Pennsylvania between April 1, 2022 and January 17, 2025
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Participant New York Heart Association (NYHA) functional class | Baseline, and at weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 108 weeks
Participant echocardiogram measurements: Left ventricular outflow tract (LVOT) gradient results at rest, Valsalva and post-exercise (if available) | Baseline, and at weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 108 weeks
Participant echocardiogram measurements: Left ventricular ejection fraction (LVEF) percentage | Baseline, and at weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 108 weeks
Participant echocardiogram measurements: Maximum left ventricular wall thickness | Baseline, and at weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 108 weeks
Participant age | Baseline
Participant gender | Baseline
Participant race | Baseline
Participant ethnicity | Baseline
Participant insurance coverage | Baseline
Participant Body Mass Index | Baseline
Participant blood pressure | Baseline
Participant heart rate | Baseline
Participant genotype | Baseline
Participant family history | Baseline
Participant New York Functional Class classification | Baseline
Participant echocardiogram measurements | Baseline
Participant comorbidities | Baseline
Participant hypertrophic cardiomyopathy (HCM) treatment history | Baseline
Mavacamten index dose prescribed | Baseline
Participant obstructive hypertrophic cardiomyopathy (oHCM) symptoms (syncope, shortness of breath, fatigue, exercise intolerance, palpitations) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts